CLINICAL TRIAL: NCT02603510
Title: A Randomized, 2X4 Week, Active-Controlled, Open-Label, 2-Treatment Arm, 2-Period Cross-Over Study Assessing the Safety of SAR342434 and Humalog® Used in Continuous Subcutaneous Insulin Infusion (CSII) in Adult Patients With Type 1 Diabetes Mellitus (T1DM)
Brief Title: Assessment of the Safety of SAR342434 and Humalog® When Administered as Continuous Subcutaneous Insulin Infusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PDY13502; U1111-1170-3739 (Other: UTN)
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — SAR342434; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAR342434/Humalog (Experimental): SAR342434 and Humalog will be self-administered subcutaneously via insulin pump. The dose will be individually titrated and administered in a basal and bolus fashion.
  Interventions: Drug: SAR342434; Drug: insulin lispro
- Humalog/SAR342434 (Experimental): Humalog and SAR342434 will be self-administered subcutaneously via insulin pump. The dose will be individually titrated and administered in a basal and bolus fashion.
  Interventions: Drug: SAR342434; Drug: insulin lispro

INTERVENTIONS:
Drug: SAR342434 — Pharmaceutical form:solution
  Route of administration: subcutaneous
Drug: insulin lispro — Pharmaceutical form:solution
  Route of administration: subcutaneous
  Other Names: Humalog

SUMMARY:
Primary Objective:

* Assess the safety of SAR342434 and Humalog when used in external pumps.

Secondary Objectives:

* Intervals for infusion set changes.
* Incidence of insulin pump alarms for infusion set occlusion.
* Patient observation of infusion set occlusion.
* Adverse events including bruising at the infusion site and injection site reactions.

DETAILED DESCRIPTION:
The study duration for each patient will be approximately 10 weeks.

ELIGIBILITY:
Inclusion criteria :

* Male and female subjects above the age of 18.
* Patients with type 1 diabetes mellitus for at least 1 year prior to the screening visit.
* At least 1 year of insulin treatment with at least 6 months of continuous subcutaneous insulin infusion (CSII) treatment with an external insulin pump.
* Signed written informed consent.

Exclusion criteria:

* HbA1c ≥8.5% at screening.
* Diabetes other than type 1 diabetes mellitus.
* History of abscess at the infusion site within 3 months prior to the screening visit (Visit 1).
* Use of oral glucose-lowering agents or any injectable glucose-lowering agents other than insulin during the 3 months before screening.
* Hospitalization for diabetic ketoacidosis (DKA) in the last 6 months before screening visit.
* Hypoglycemic unawareness as judged by the Investigator in the last 6 months before the screening visit.
* History of severe hypoglycemia requiring treatment by emergency room admission or hospitalization in the last 6 months before screening visit.
* Any clinically significant abnormality identified on physical examination, laboratory tests, or vital signs at the time of screening that in the judgment of the investigator or any sub investigator would preclude safe completion of the study.
* Known history of drug or alcohol abuse within 6 months prior to the time of screening.
* Use of investigational drug(s) within 3 months or 5 half-lives, whichever is longer, prior to the screening visit.
* Patients who had previously received SAR342434 in any other clinical trial.
* Pregnancy and lactation: Women of child bearing potential (WOCPB) (premenopausal, not surgically sterile for at least 3 months prior to the time of screening) not using highly effective (ie, with low failure rate <1% per year) method(s) of birth control throughout the study and/or unwilling to be tested for pregnancy.
* Any contraindication to the use of Humalog as defined in the national product labels; history of hypersensitivity to Humalog or to any of the excipients.
* Patients is an employee or relative of an employee of the Sponsor.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Frequency of infusion set occlusions | 4 weeks

SECONDARY OUTCOMES:
Number of infusion set changes in each treatment period | 4 weeks
Number of insulin pump alarms for infusion set occlusions | 4 weeks
Number of adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- United States (2):
  - Investigational Site Number 840002, Little Rock, Arkansas
  - Investigational Site Number 840001, Denver, Colorado

REFERENCES:
- [Derived] Thrasher J, Surks H, Nowotny I, Pierre S, Rotthaeuser B, Wernicke-Panten K, Garg S. Safety of Insulin Lispro and a Biosimilar Insulin Lispro When Administered Through an Insulin Pump. J Diabetes Sci Technol. 2018 May;12(3):680-686. doi: 10.1177/1932296817753644. Epub 2018 Jan 23. PMID 29359575